CLINICAL TRIAL: NCT01901874
Title: GORE® Carotid Stent Clinical Study for the Treatment of Carotid Artery Stenosis in Patients at Increased Risk for Adverse Events From Carotid Endarterectomy
Brief Title: The Gore SCAFFOLD Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCS 10-08
Record Dates: First submitted 2013-07-12; First posted 2013-07-17 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Carotid Artery Disease; Carotid Artery Stenosis
Keywords: Stroke; Carotid Artery Stenting (CAS); Embolic Protection Device (EPD); Stent; Carotid Stenosis; Constriction, Pathologic; Carotid Artery Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Pathological Conditions, Anatomical; Angioplasty
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke; Constriction, Pathologic; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Arterial Occlusive Diseases; Vascular Diseases; Cardiovascular Diseases; Pathological Conditions, Anatomical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carotid Artery Stenting (Experimental): Carotid Artery Stenting with the GORE® Carotid Stent
  Interventions: Device: Carotid Artery Stenting

INTERVENTIONS:
Device: Carotid Artery Stenting — Carotid Artery Stenting with the GORE® Carotid Stent
  Other Names: GORE® Carotid Stent

SUMMARY:
Evaluate the safety and efficacy of the GORE® Carotid Stent for the treatment of carotid artery stenosis in patients at increased risk for adverse events from carotid endarterectomy

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-arm clinical study comparing outcomes with the GORE® Carotid Stent to a performance goal derived from carotid endarterectomy outcomes in high-surgical-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years old at informed consent
* Patient is willing and capable of complying with all study protocol requirements, including specified follow-up period and can be contacted by telephone.
* Patient is willing to provide written informed consent prior to enrollment in study.
* Patient is either:

  * Symptomatic with carotid stenosis ≥50% as determined by angiography using NASCET methodology. Symptomatic is defined as amaurosis fugax ipsilateral to the carotid lesion; Transient Ischemic Attack (TIA) or non-disabling stroke within 180 days of the procedure within the hemisphere supplied by the target vessel; OR
  * Asymptomatic with carotid stenosis ≥80% as determined by angiography using NASCET methodology
* Patient must be considered high risk for adverse events during carotid endarterectomy

Note: Additional inclusion criteria may apply

Exclusion Criteria:

* Patient has life expectancy of less than one year.
* Patient is experiencing (or has experienced) an evolving, acute, or recent disabling stroke.
* Patient has anticipated or potential sources of emboli (e.g. atrial fibrillation, known previously symptomatic patent foramen ovale (PFO), mechanical heart valve, or Deep Vein Thrombosis (DVT) treated within 6 months).
* Patient has had an acute myocardial infarction within 72 hours prior to the index procedure.
* Patient has a history of major, disabling ipsilateral stroke with residual deficit that may confound the neurological subject assessments.
* Patient has known severe carotid stenosis contralateral to the target lesion requiring treatment within 30 days following the index procedure.

Note: Additional exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Lankenau Heart Institute; Peter Schneider, MD, Principal Investigator — Kaiser Health System, Honolulu
Locations (2):
- United States (2):
  - Kaiser Permanente Hawaii, Honolulu, Hawaii
  - Lankenau Heart Institute, Wynnewood, Pennsylvania

REFERENCES:
- [Derived] Gray WA, Levy E, Bacharach JM, Metzger DC, Randall B, Siddiqui A, Schonholz C, Alani F, Schneider PA. Evaluation of a novel mesh-covered stent for treatment of carotid stenosis in patients at high risk for endarterectomy: 1-year results of the SCAFFOLD trial. Catheter Cardiovasc Interv. 2020 Jul;96(1):121-127. doi: 10.1002/ccd.28586. Epub 2019 Nov 11. PMID 31713310

RESULTS

PARTICIPANT FLOW:
Period: Procedure
Arm/Group | Carotid Artery Stenting
Started | 312
Completed | 312
Not Completed | 0
Period: Screening Committee Retrospective Review
Arm/Group | Carotid Artery Stenting
Started | 312
Completed | 265
Not Completed | 47
Not completed — Protocol Violation | 47
Period: 30-Day MAE Evaluation
Arm/Group | Carotid Artery Stenting
Started | 265
Completed | 264
Not Completed | 1
Not completed — Insufficient Follow-up | 1
Period: 1-Year (365-Day) MAE Evaluation
Arm/Group | Carotid Artery Stenting
Started | 264
Completed | 244
Not Completed | 20
Not completed — Death | 7
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 2
Not completed — Insufficient Follow-up | 6

BASELINE CHARACTERISTICS:
Population: Per protocol subjects
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 265
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.1 (8.8)
Age, Continuous [Median (Full Range); unit: years] | 74.4 [45.8 to 92.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 258
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 252
  More than one race | 3
  Unknown or Not Reported | 0
Diabetes Mellitus [Count of Participants; unit: Participants] | 107
Hypertension [Count of Participants; unit: Participants] | 249
Cigarette Smoking [Count of Participants; unit: Participants]
  Current or stopped <12 months ago | 67
  Previous (stopped >12 months ago) | 139
  Never | 59
Previous Carotid Disease [Count of Participants; unit: Participants] | 125
Symptomatic [Count of Participants; unit: Participants] | 33
History of Ischemic Stroke [Count of Participants; unit: Participants] | 48
History of Transient Ischemic Attack (TIA) [Count of Participants; unit: Participants] | 40
Ipsilateral Amaurosis Fugax or Transient Monocular Blindness (TMB) [Count of Participants; unit: Participants] | 9
Endarterectomy [Count of Participants; unit: Participants] | 79
Target Lesion Location [Count of Participants; unit: Participants]
  ICA | 235
  Bifurcation | 30
Target Vessel Reference Diameter (mm) [Median (Full Range); unit: millimeters] | 5.5 [3.7 to 9.0]
Target Lesion Length (mm) [Median (Full Range); unit: millimeters] | 20 [1 to 40]
Target Lesion % Diameter Stenosis [Median (Full Range); unit: percentage of vessel diameter] — = (RVD - MLD) / RVD x 100, where RVD = Reference Vessel Diameter (mm) and MLD = Minimum Lumen Diameter (mm)
  percentage of vessel diameter | 85 [50 to 99]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Major Adverse Events (MAE) at One Year
Description: MAE defined as any death, stroke, or myocardial infarction through 30 days post-index procedure, or ipsilateral stroke between 31 days and 1 year (365 days).
Time Frame: 365 days
Population: Per protocol subjects with 1-year MAE evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 244
Participants | 11
Statistical Analysis 1: Comparison: Carotid Artery Stenting; Test null hypothesis of equal or greater proportion with 1-year MAE compared to a performance goal (PG). H0: P ≥ 16.9% vs H1: P < 16.9%, where P is the true proportion of CAS subjects with 1-year MAE and 16.9% is the PG based on outcomes reported for patients treated with carotid endarterectomy (CEA). N=280 subjects provide ≥90% power to exclude PG with 95.1% confidence if P=10.2% under H1; Test type: Other — Acceptable performance: favorably exclude PG=16.9% with 95.1% confidence. Wa = expected weight (proportion) anatomic = 35% Pa = CEA expected anatomic MAE = 11% Wc = expected weight (proportion) comorbid = 65% Pc = CEA expected comorbid MAE = 14% D = noninferiority delta = 4% PG = 0.35 x 11% + 0.65 x 14% + 4% = 16.9%; p < 0.00001, Binomial test (normal approximation) — A priori 1-sided alpha = 0.049 (from simulation) to ensure overall type-1 error rate ≤ 0.05; Weighted binomial proportion = 0.0448, 95.1% CI 1-sided [upper limit 0.0846], Standard Error of Mean 0.0241 — Weighted by expected fractions of anatomic and comorbid high risk subjects (35% and 65%, respectively). Standard error based on H0

2. Secondary Outcome: Number of Participants Who Achieved Stent Technical Success
Description: Stent Technical Success defined as successful implantation of a GORE® Carotid Stent
Time Frame: Procedural
Population: Per protocol subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 265
Participants | 265

3. Secondary Outcome: Number of Participants Who Achieved Embolic Protection Device (EPD) Technical Success
Description: EPD Technical Success defined as GORE® Embolic Filter delivered, placed, and retrieved without requiring assisting interventional methods.
Time Frame: Procedural
Population: Per protocol subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 265
Participants | 251

4. Secondary Outcome: Number of Participants Who Achieved Procedure Success
Description: Procedure Success defined as Stent Technical Success with < 30% residual stenosis and no in-hospital MAE.
Time Frame: Procedural
Population: Per protocol subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 265
Participants | 250

5. Secondary Outcome: Number of Participants Who Experienced MAE at 30 Days
Description: Defined as any death, stroke, or myocardial infarction through 30 days post-index procedure.
Time Frame: 30 days
Population: Per protocol subjects with 30-day MAE evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 264
Participants | 8

6. Secondary Outcome: 30-Day MAE - Death
Description: Any cause death through 30 days post-index procedure
Time Frame: 30 days
Population: Per protocol subjects with 30-day MAE evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 264
Participants | 1

7. Secondary Outcome: 30-Day MAE - Myocardial Infarction
Description: Any myocardial infarction through 30 days post-index procedure
Time Frame: 30 days
Population: Per protocol subjects with 30-day MAE evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 264
Participants | 4

8. Secondary Outcome: 30-Day MAE - Stroke
Description: Any stroke through 30 days post-index procedure
Time Frame: 30 days
Population: Per protocol subjects with 30-day MAE evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 264
Participants | 3

9. Secondary Outcome: In-Stent Restenosis
Description: ≥80% diameter stenosis within the stented lesion or within 5 mm proximal or distal to the stent at follow-up evaluation by core lab angiographic analysis
Time Frame: 365 days
Population: Per protocol subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 265
Participants | 4
Statistical Analysis 1: Comparison: Carotid Artery Stenting; Test type: Other; Cumulative probability = 0.018, 95% CI 2-sided [0.007 to 0.047] — Kaplan-Meier product-limit method (Greenwood's formula for standard error)

10. Secondary Outcome: Target Lesion Revascularization
Description: Any clinically driven revascularization procedure that is performed to increase the luminal diameter inside or within 5 mm of the previously treated lesion
Time Frame: 365 days
Population: Per protocol subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Carotid Artery Stenting
Number analyzed (Participants) | 265
Participants | 5
Statistical Analysis 1: Comparison: Carotid Artery Stenting; Test type: Other; Cumulative probability = 0.022, 95% CI 2-sided [0.009 to 0.052] — Kaplan-Meier product-limit method (Greenwood's formula for standard error)

ADVERSE EVENTS:
Time Frame: 395 days (end of 1-year follow-up window)
Arm/Group | Carotid Artery Stenting
All-Cause Mortality (participants affected / at risk) | 11/265
Serious Adverse Events (participants affected / at risk) | 104/265
Other Adverse Events (participants affected / at risk) | 110/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotid Artery Stenting (N=265)
Anaemia (Blood and lymphatic system disorders) | 4 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 4 (4)
Angina pectoris (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 5 (5)
Left ventricular failure (Cardiac disorders) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 (4)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2)
Vascular stent restenosis (General disorders) | 10 (11)
Vascular stent thrombosis (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 10 (10)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Autonomic dysreflexia (Injury, poisoning and procedural complications) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (2)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Adenosquamous cell lung cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Carotid artery dissection (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 9 (9)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 6 (6)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (2)
Hypoaesthesia (Nervous system disorders) | 1 (2)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Device breakage (Product Issues) | 1 (1)
Device malfunction (Product Issues) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Aortic aneurysm (Vascular disorders) | 3 (3)
Aortic aneurysm rupture (Vascular disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 9 (10)
Intermittent claudication (Vascular disorders) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Subclavian artery thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carotid Artery Stenting (N=265)
Anaemia (Blood and lymphatic system disorders) | 6 (6)
Angina pectoris (Cardiac disorders) | 5 (5)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 9 (10)
Constipation (Gastrointestinal disorders) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 6 (6)
Peripheral swelling (General disorders) | 4 (4)
Bronchitis (Infections and infestations) | 4 (4)
Influenza (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 4 (4)
Urinary tract infection (Infections and infestations) | 14 (16)
Incision site haematoma (Injury, poisoning and procedural complications) | 5 (5)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 8 (8)
Laceration (Injury, poisoning and procedural complications) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5)
Dizziness (Nervous system disorders) | 8 (8)
Headache (Nervous system disorders) | 14 (16)
Hypoaesthesia (Nervous system disorders) | 4 (4)
Syncope (Nervous system disorders) | 5 (5)
Mental status changes (Psychiatric disorders) | 3 (3)
Urinary retention (Renal and urinary disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Haematoma (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 9 (9)
Hypotension (Vascular disorders) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2014-10-22): https://cdn.clinicaltrials.gov/large-docs/74/NCT01901874/Prot_000.pdf
  • Statistical Analysis Plan (2014-06-10): https://cdn.clinicaltrials.gov/large-docs/74/NCT01901874/SAP_001.pdf